CLINICAL TRIAL: NCT04956835
Title: The Implementation of the Classification of Intraoperative Adverse Events (ClassIntra) for Neurosurgical Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Richard Drexler, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: CINS
Record Dates: First submitted 2021-06-26; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Neurological Morbidity; Surgical Complication; Anesthesia Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the planned study, the ClassIntra score will be assessed after all neurosurgical procedures in the upcoming 6 months and correlated with all pre- and postoperative data. Afterwards, the conclusion will be made, if the ClassIntra score could predict the postoperative course of the patients regarding their neurological and general condition. Furthermore, analyses will be made to develop novel postoperative routines adjusted to the individual ClassIntra score of the patient.

DETAILED DESCRIPTION:
Surgeons strive for the best possible outcome of their surgeries with the greatest possible chance for recovery of the patients. Therefore, monitoring and quality improvement is increasingly important in surgery. As there are well-defined scores and classifications to describe the postoperative course regarding morbidity, mortality and neurological status, no validated classification for intraoperative quality exists by now. However, Dell-Kuster et al. introduced a novel classification for assessing all intraoperative adverse events: ClassIntra. This classification was developed in a Delphi consensus containing international, interdisciplinary, and validated in a multicentre cohort study across all surgical disciplines. The classification defines intraoperative adverse events as any deviation from the ideal intraoperative course occurring between skin incision and skin closure and contains any event related to surgery and anaesthesia. Depending on the kind of adverse event, the ClassIntra score ranges from 0 (no event) to 5 (intraoperative death). A prospective study with a main focus on neurosurgery covering the whole spectrum of elective and emergency procedures is needed. Hereby, the outcome parameters need to be defined specific for neurosurgical procedures including a preoperative and postoperative neurological status.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery at a neurosurgical department

Exclusion Criteria:

* Patients under 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery at a neurosurgical department either elective or emergency surgery
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications according to Clavien-Dindo classification | within two weeks after surgery
  Grade 0 to V (0 no complication, V death)
Comprehensive Complication Index | within two weeks after surgery
  Based on Clavien-Dindo classification with a scale from 0 to 100 (0 no complication, 100 death)
Neurological status | within two weeks after surgery
  classified to NANO scale, NIHSS, modified Rankin Scale, Glasgow Outcome Scale
Neurological outcome (NANO scale) | within two weeks after surgery
  according to neurological assessment in neuro-oncology (NANO) with a scale from 0 to 23 (0 no neurological deficit, 23 multiple neurological deficits)
Neurological outcome (NIHSS) | within two weeks after surgery
  according to National Institutes of Health Stroke Scale (0 no stroke symptoms 1-4 minor stroke 5-15 moderate stroke 16-20 moderate to severe stroke 21-42 severe stroke)
Neurological outcome (mRS) | within two weeks after surgery
  according to modified Rankin Scale with a scale from 0 to 6 (0 no symptoms, 6 dead)
In-hospital mortality | within two weeks after surgery
  Death of the patient

SECONDARY OUTCOMES:
Length of ICU stay | within two weeks after surgery
Length of hospital stay | within two weeks after surgery
Readmission rate | within 90 days after surgery
  Readmission to hospital after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Richard Drexler, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hambrug, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dell-Kuster S, Gomes NV, Gawria L, Aghlmandi S, Aduse-Poku M, Bissett I, Blanc C, Brandt C, Ten Broek RB, Bruppacher HR, Clancy C, Delrio P, Espin E, Galanos-Demiris K, Gecim IE, Ghaffari S, Gie O, Goebel B, Hahnloser D, Herbst F, Ioannidis O, Joller S, Kang S, Martin R, Mayr J, Meier S, Murugesan J, Nally D, Ozcelik M, Pace U, Passeri M, Rabanser S, Ranter B, Rega D, Ridgway PF, Rosman C, Schmid R, Schumacher P, Solis-Pena A, Villarino L, Vrochides D, Engel A, O'Grady G, Loveday B, Steiner LA, Van Goor H, Bucher HC, Clavien PA, Kirchhoff P, Rosenthal R. Prospective validation of classification of intraoperative adverse events (ClassIntra): international, multicentre cohort study. BMJ. 2020 Aug 25;370:m2917. doi: 10.1136/bmj.m2917. PMID 32843333
- [Derived] Drexler R, Ricklefs FL, Pantel T, Gottsche J, Nitzschke R, Zollner C, Westphal M, Duhrsen L. Association of the classification of intraoperative adverse events (ClassIntra) with complications and neurological outcome after neurosurgical procedures: a prospective cohort study. Acta Neurochir (Wien). 2023 Aug;165(8):2015-2027. doi: 10.1007/s00701-023-05672-w. Epub 2023 Jul 5. PMID 37407852